CLINICAL TRIAL: NCT01305824
Title: Multicenter, Double-Blind, Placebo-Controlled Study of PRT-201 Administered Immediately After Arteriovenous Fistula Creation in Patients With Chronic Kidney Disease
Brief Title: A Study of PRT-201 Administered Immediately After Arteriovenous Fistula Creation in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT-201-201
Record Dates: First submitted 2011-02-16; First posted 2011-03-01 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease
Keywords: arteriovenous fistula; AVF; hemodialysis; vascular access; dialysis; fistula; PRT-201; vonapanitase; kidney; renal
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Fistula | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRT 201 (10 micrograms) (Active Comparator)
  Interventions: Drug: PRT-201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PRT-201 (30 micrograms) (Active Comparator)
  Interventions: Drug: PRT-201

INTERVENTIONS:
Drug: PRT-201 — PRT-201 10 micrograms administered at the time of AVF creation.
  Arms: PRT 201 (10 micrograms)
Drug: Placebo — Placebo administered at the time of AVF creation.
  Arms: Placebo
Drug: PRT-201 — PRT-201 30 micrograms administered at the time of AVF creation.
  Arms: PRT-201 (30 micrograms)

SUMMARY:
The purpose of this study is to determine if PRT-201 when applied to a limited segment of your blood vessel (about 2 inches) immediately after surgery to create an arteriovenous fistula is safe and improves the patency of your fistula. PRT-201 is a protein that has been shown to help keep vessels open ("patent") when applied to the outside surface of the blood vessels (arteries and veins) in AVF patients in a previous study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Life expectancy of at least 6 months.
3. Chronic kidney disease on hemodialysis, or with anticipated start of hemodialysis within 6 months.
4. Planned creation of a new radiocephalic or brachiocephalic AVF. Revisions of an existing AVF and transposed AVF are not acceptable.

Exclusion Criteria:

1. History or presence of an arterial aneurysm.
2. Malignancy or treatment for malignancy within the previous 12 months with the exception of the following cancers if they have been resected: localized basal cell cancer, squamous cell skin cancer, or any cancer in situ.
3. Hepatic dysfunction defined as bilirubin, ALT [SGPT] or AST [SGOT] >2.5 times the upper limit of normal, decompensated cirrhosis, ascites, or known esophageal or gastric varices.
4. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within 90 days prior to signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Primary AVF patency. | 12 months after AVF creation
Number of participants with adverse events as a measure of safety and tolerability of PRT-201. | 12 months after AVF creation.

SECONDARY OUTCOMES:
Secondary Fistula Patency | 12 months after AVF creation

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - California Institute of Renal Research, San Diego, California
  - Kaiser Permanente, San Diego, California
  - UCSF, San Francisco, California
  - Rush Medical Center, Chicago, Illinois
  - Renal Care Associates, Peoria, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Vascular Specialty Center, Baton Rouge, Louisiana
  - Beth Israel Deconness Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMASS Medical Center, Worcester, Massachusetts
  - St Clair Specialty Physicians, Detroit, Michigan
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Legacy Oregon Surgical, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia

REFERENCES:
- [Result] Hye RJ, Peden EK, O'Connor TP, Browne BJ, Dixon BS, Schanzer AS, Jensik SC, Dember LM, Jaff MR, Burke SK. Human type I pancreatic elastase treatment of arteriovenous fistulas in patients with chronic kidney disease. J Vasc Surg. 2014 Aug;60(2):454-461.e1. doi: 10.1016/j.jvs.2014.02.037. Epub 2014 Mar 27. PMID 24684771